CLINICAL TRIAL: NCT02681445
Title: Non-invasive TB Triage and Patient Mapping Platform Using Breath Via Low-Cost Titanium Dioxide Nanotube Sensor
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Swomitra Mohanty, Assistant Professor, University of Utah
Other Study IDs: 00088349
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Group 1 Healthy Non Smokers: No TB Symptoms No TB History Negative Mantoux test Normal Chest X-ray Non-Smoker
  Interventions: Device: Breath Collection
- Group-2 Smokers: No TB History No TB Symptoms No TB History Negative Mantoux test Smoker 10 + Cigarettes/day
  Interventions: Device: Breath Collection
- HIV Positive: No TB Symptoms No TB History Negative Mantoux test Normal Chest X-ray HIV Positive
  CD4 count >200
  Interventions: Device: Breath Collection
- TB Suspect Group: WHO Screening Recommendation Protocls Unexplained Cough Sputum production Fever Weight Loss or loss of appetite Night Sweats
  Interventions: Device: Breath Collection
- Lower Respiratory Track Infection: TB Lab test Negative Ab Normal Chest X-ray HIV Negative
  Interventions: Device: Breath Collection

INTERVENTIONS:
Device: Breath Collection — breath will be collected from patients in breath bag for analysis for observational study.

SUMMARY:
The purpose of this pilot study is to evaluate the sensitivity and specificity of a nanotube-based point-of-care breath-based tuberculosis screening test as compared to the current standards of care including sputum microscopy, sputum culture, chest X-ray, and GeneXpert (MTB/RIF).

The primary objective is to determine an initial estimate of the sensitivity and specificity of a nano-tube based point-of-care test for the diagnosis and screening of active pulmonary tuberculosis.

Secondary objectives include the collection of user data to test and further develop the screening platform based on end-user feedback.

DETAILED DESCRIPTION:
TB is an infectious disease caused by various strains of mycobacteria. It typically infects the lungs and is spread through the air when an infected patient sneezes, coughs, or spits. When this occurs, the TB bacilli are propelled into the air in droplets that can remain suspended for long periods of time. An individual simply needs to inhale a small amount of bacilli to become infected.

Conventional methods for TB detection and diagnosis are traditionally performed in laboratories or hospitals. For example, the most common method for diagnosis of TB is the acid fast staining of a sputum sample which is then followed by a sputum smear microscopy test. However a disadvantage with the sputum smear test is its poor sensitivity, which is estimated to be at 70%. Additionally, the sensitivity of sputum smear spectroscopy in field settings has been shown to be much lower (35%), especially in populations that have high rates of TB and HIV coinfection. Culturing of mycobacterium from sputum samples is a more sensitive technique. Sputum samples are collected and cultured in either solid media or liquid media looking for the presence of the mycobacterium. However this methodology takes time to conduct (3-4 weeks for solid cultures, and 10-14 days for liquid cultures), which makes it difficult to employ in low resource settings that are typically far from testing facilities.

Recently, other technologies have been developed including fluorescence microscopy for smear tests (10% more sensitive than light microscopy), LED fluorescent microscopy for inexpensive imaging equipment that can be used in the field without the need for a darkroom, and rapid culturing techniques to reduce incubation time. Despite all the improvements that have been made in TB diagnosis, no simple inexpensive POC test is currently available. The techniques mentioned above either focus on variations of microscopy or culture technique. In either case, these methods require lab facilities and highly trained personnel that typically are not available in many rural or low resource areas.

Recent research has shown that various strains of the mycobacteria produce distinct gaseous volatile biomarkers that can be used as a methodology for detecting and identifying the mycobacterium. Specifically, Syhre and Chambers found that Mycobacterium tuberculosis and Mycobacterium bovis cultures give off four specific volatile organic biomarkers (VOBs): methyl phenylacetate, methyl p-anisate, methyl nicotinate, and o-phenylanisole. These compounds were detectable before the visual appearance of colonies, which could have implications in detection of latent TB infection. Syhre et al. were able to detect statistically significant differences of methyl nicotinate in the breath of smear positive TB patients when compared to healthy (smear negative) subjects. Analyses in these studies were done using gas chromatography/mass spectroscopy analysis tools. While they are effective in identifying and quantifying complex gas samples, they are expensive, bulky, and not appropriate for point of care (POC) diagnostics.

These challenges associated with the diagnosis of TB are significant as TB is the second leading cause of death due to a single infectious organism and is responsible for 1.3 million deaths annually (over 3,500 every day), according to the WHO. Overall, an estimated 2 billion people are currently infected worldwide with 8.6 million new active infections occurring each year.[8] Each of these individuals can transmit the disease to 10 to 15 people per year and face a mortality rate of 50% if untreated. The economic burden of TB is staggering as the World Bank estimates that high burden countries can lose up to 7% of GDP due to productivity losses from TB patients and their caretakers. It is so critical that the World Bank committed $100 million to testing for and treating TB in India in 2014 alone.

Of the 8.6 million new active TB cases that occur annually, the WHO estimates that roughly 3 million of these patients are 'missed' and do not receive the diagnosis or care they need. One of the primary reasons for this gap is delays in accessing TB-related care or long lead times for diagnostic tests. As a result, developing new large scale screening tests (also known as triage or 'rule out' tests) are particularly needed due to the fact that up to 80% of people tested for TB do not have active disease, stretching the limited and valuable resources that are devoted for diagnostic testing. As a result, FIND, a world leader in guiding and coordinating research and development for diseases such as TB, ranked the development of new screening tests as one of the top 3 priorities in the fight against TB.

This pilot study will be conducted to determine if a newly developed sensing methodology for screening TB at the POC based on volatile biomarkers is feasible through the use of a low cost solid-state sensor using functionalized 3D TiO2 nanotube arrays that bind the volatile biomarkers. If the clinical sensitivity is sufficient, this technology could provide a means for identifying many of the 'missed' TB patients and allow testing resources and efforts to be focused on those at the highest risk of having the disease.

Previously, we have tested the breath profile of a small number patients from local TB clinics and have confirmed the presence of these biomarkers in their breath (IRB_0065207). Larger patients studies are now required to gain an estimate of the sensitivity and specificity to determine the potential of using the sensor as a screening test. This study will be conducted in Mumbai, India with the University's Research Electronic Data Capture (REDCap) system used to securely collect and store the data from this study.

This study has been reviewed and approved by the Mahatma Gandhi Mission Institute of Health Sciences Ethical Committee for Research on Human Subjects and Scientific Advisory Committee.

ELIGIBILITY:
Inclusion Criteria:

* No TB Symtoms No history of TB Negative Mantoux test Normal Chest X-ray HIV Negative

Exclusion Criteria:

Prior history of TB

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study type: Observational feasibility study
  * Study population: Non-pregnant adults over the age of 18 from the areas around Mumbai, India. Based upon records of these clinical sites, about 5% to 7% of the patients reporting at these hospitals are suspected to be TB positive.
  * Endpoint: Estimate of the diagnostic accuracy of a POC TB biomarker breath test (sensitivity, specificity).
  * Phase: Phase I (feasibility or pilot study)
  * Study sites: Multicenter trial (4 clinical sites in Mumbai, India)
  * Study groups: 5
  * Sample Size (approx): 800
  * Estimated enrollment time: 1 year
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Correlation of sensor ability to detect breath biomarkers for TB | 12 Months
  Assess feasability of TB sensor to detect breath biomarkers from patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahatma Gandhi Institute of Health Science, Navi Mumbai, India